CLINICAL TRIAL: NCT03487861
Title: Development of a Diagnostic Kit for Urinary Transglutaminase 2 as a Biomarker for Kidney Allograft Fibrosis
Brief Title: Urinary Transglutaminase 2 as a Biomarker for Kidney Allograft Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung Shin, Associate professor, Asan Medical Center
Other Study IDs: NRF-2016M3A9E8941330
Record Dates: First submitted 2018-03-18; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Kidney Allograft Fibrosis; Kidney Transplant Failure and Rejection
Keywords: transglutaminase type 2; kidney transplantation; chronic allograft nephropathy; biomarker
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: observational(urinary biomarker for kidney allograft fibrosis) — After an informed consent is obtained, urine specimens will be collected prospectively before kidney transplantation (if available) and 3rd and 7th day, 1st, 3rd, and 6th month post-transplant. About 35~50ml of urine sample is collected from each patient. For each urine specimen, 0.5 ml of a protease inhibitor mixture (5mM 4-(2-animoethyl) benzensulfonyl fluoride hydrolchloride, 2 μM Leupeptin-hemisulfate, and 3.3 mM Sodium azide) is added. To remove urinary sediments including whole cells, large membrane particles, and other debris, urine specimens are centrifuged at a rate of 4000 rpm for 15 minutes at 4 ℃. An aliquot of supernatant is stored at -80 ℃ until use. Urinary biomarkers including transglutaminase 2 are quantified using ELISA or CBA. In addition, urinary exosomes are isolated and analyzed. When a for-cause biopsy is done for some patients, the correlation between biomarkers and pathologic diagnosis will be assessed.

SUMMARY:
The aim of this study is to verify the ability of transglutaminase type 2 to predict rejection or chronic allograft nephropathy of renal allograft. On the basis of biomolecular mechanisms aggravating chronic allograft nephropathy, we eventually expect to develop the remedy to prevent chronic allograft nephropathy after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients from cadaveric or living donors
* kidney transplant recipients who take immunosuppressants regularly
* kidney transplant recipients who voluntarily agree to participate in this trial

Exclusion Criteria:

* multiorgan transplant recipients
* kidney transplant recipients with active infection
* kidney transplant recipients with alcohol or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney transplant recipients from cadaveric or living donors
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change of level of urinary transglutaminase 2 | 3 days, 7 days, 1 month, 3 months, 6 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: SUNG SHIN, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Meguid El Nahas A, Bello AK. Chronic kidney disease: the global challenge. Lancet. 2005 Jan 22-28;365(9456):331-40. doi: 10.1016/S0140-6736(05)17789-7. PMID 15664230
- [Result] Lorand L, Graham RM. Transglutaminases: crosslinking enzymes with pleiotropic functions. Nat Rev Mol Cell Biol. 2003 Feb;4(2):140-56. doi: 10.1038/nrm1014. PMID 12563291
- [Result] Oh K, Park HB, Byoun OJ, Shin DM, Jeong EM, Kim YW, Kim YS, Melino G, Kim IG, Lee DS. Epithelial transglutaminase 2 is needed for T cell interleukin-17 production and subsequent pulmonary inflammation and fibrosis in bleomycin-treated mice. J Exp Med. 2011 Aug 1;208(8):1707-19. doi: 10.1084/jem.20101457. Epub 2011 Jul 11. PMID 21746810
- [Result] Kojima S, Nara K, Rifkin DB. Requirement for transglutaminase in the activation of latent transforming growth factor-beta in bovine endothelial cells. J Cell Biol. 1993 Apr;121(2):439-48. doi: 10.1083/jcb.121.2.439. PMID 8096847
- [Result] Scarpellini A, Germack R, Lortat-Jacob H, Muramatsu T, Billett E, Johnson T, Verderio EA. Heparan sulfate proteoglycans are receptors for the cell-surface trafficking and biological activity of transglutaminase-2. J Biol Chem. 2009 Jul 3;284(27):18411-23. doi: 10.1074/jbc.M109.012948. Epub 2009 Apr 27. PMID 19398782
- [Result] Scarpellini A, Huang L, Burhan I, Schroeder N, Funck M, Johnson TS, Verderio EA. Syndecan-4 knockout leads to reduced extracellular transglutaminase-2 and protects against tubulointerstitial fibrosis. J Am Soc Nephrol. 2014 May;25(5):1013-27. doi: 10.1681/ASN.2013050563. Epub 2013 Dec 19. PMID 24357671
- [Result] Melhem A, Muhanna N, Bishara A, Alvarez CE, Ilan Y, Bishara T, Horani A, Nassar M, Friedman SL, Safadi R. Anti-fibrotic activity of NK cells in experimental liver injury through killing of activated HSC. J Hepatol. 2006 Jul;45(1):60-71. doi: 10.1016/j.jhep.2005.12.025. Epub 2006 Feb 8. PMID 16515819
- [Result] Shin S, Kim YH, Cho YM, Park Y, Han S, Choi BH, Choi JY, Han DJ. Interpreting CD56+ and CD163+ infiltrates in early versus late renal transplant biopsies. Am J Nephrol. 2015;41(4-5):362-9. doi: 10.1159/000430473. Epub 2015 Jun 18. PMID 26087825
- [Result] Victorino F, Sojka DK, Brodsky KS, McNamee EN, Masterson JC, Homann D, Yokoyama WM, Eltzschig HK, Clambey ET. Tissue-Resident NK Cells Mediate Ischemic Kidney Injury and Are Not Depleted by Anti-Asialo-GM1 Antibody. J Immunol. 2015 Nov 15;195(10):4973-85. doi: 10.4049/jimmunol.1500651. Epub 2015 Oct 9. PMID 26453755
- [Result] Brusilovsky M, Radinsky O, Cohen L, Yossef R, Shemesh A, Braiman A, Mandelboim O, Campbell KS, Porgador A. Regulation of natural cytotoxicity receptors by heparan sulfate proteoglycans in -cis: A lesson from NKp44. Eur J Immunol. 2015 Apr;45(4):1180-91. doi: 10.1002/eji.201445177. Epub 2015 Jan 21. PMID 25546090
- [Result] Breggia AC, Himmelfarb J. Primary mouse renal tubular epithelial cells have variable injury tolerance to ischemic and chemical mediators of oxidative stress. Oxid Med Cell Longev. 2008 Oct-Dec;1(1):33-8. doi: 10.4161/oxim.1.1.6491. PMID 19794906
- [Result] Jeong EM, Kim CW, Cho SY, Jang GY, Shin DM, Jeon JH, Kim IG. Degradation of transglutaminase 2 by calcium-mediated ubiquitination responding to high oxidative stress. FEBS Lett. 2009 Feb 18;583(4):648-54. doi: 10.1016/j.febslet.2009.01.032. Epub 2009 Feb 1. PMID 19183553
- [Result] Anglicheau D, Muthukumar T, Hummel A, Ding R, Sharma VK, Dadhania D, Seshan SV, Schwartz JE, Suthanthiran M. Discovery and validation of a molecular signature for the noninvasive diagnosis of human renal allograft fibrosis. Transplantation. 2012 Jun 15;93(11):1136-46. doi: 10.1097/TP.0b013e31824ef181. PMID 22592886
- [Result] Halloran PF, Famulski KS, Reeve J. Molecular assessment of disease states in kidney transplant biopsy samples. Nat Rev Nephrol. 2016 Sep;12(9):534-48. doi: 10.1038/nrneph.2016.85. Epub 2016 Jun 27. PMID 27345248